CLINICAL TRIAL: NCT04167371
Title: Treament of Rumination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)373/2019
Record Dates: First submitted 2019-11-15; First posted 2019-11-18 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2020-12

CONDITIONS: Rumination Disorders
MeSH Terms: conditions — Rumination Syndrome | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback (Experimental)
  Interventions: Behavioral: Biofeedback
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Behavioral: Biofeedback — Three sessions by biofeedback will be performed during the first 3 weeks of the intervention period. In each session patients will be taught to control abdominal and thoracic muscular activity by providing a visual display of the abdominal and thoracic perimeter; patients will be instructed to perform the same exercises before and after breakfast, lunch and dinner during the 4-week intervention period.
  Arms: Biofeedback
Dietary Supplement: Placebo — Three sessions will be performed during the first 3 weeks of the intervention period. In each session abdominal and thoracic perimeter will be recorded but not shown to the patient; patients will take a pill of placebo containing 0.5 g glucose and no specific instructions will be provided. Patients will be instructed to take a pill of placebo before breakfast, lunch and dinner during the 4-week intervention period.
  Arms: Placebo

SUMMARY:
Background. Rumination syndrome is characterized by effortless recurrent regurgitation of recently ingested food into the mouth, with consequent expulsion or re-chewing and swallowing. In a previous study we showed that rumination is produced by an unperceived, somatic response to food ingestion. We developed an original biofeedback technique based on electromyography-guided control of abdominothoracic muscular activity. In a randomized, placebo-controlled trial we demonstrated the superiority of biofeedback over placebo for the treatment of rumination. However, the technique is technically complex and unpractical.

Aim. To prove the efficacy of a simplified biofeedback technique for the treatment of rumination. Selection criteria. Rumination after meal ingestion. Intervention. Patients will be randomized into biofeedback in placebo groups. Three sessions of either biofeedback or placebo intervention will be performed after ingestion of a probe meal during the first 3 weeks of the 4 weeks intervention period.

Biofeedback: patients will be taught to control abdominal and thoracic muscular activity by providing a visual display of the abdominal and thoracic perimeter; patients will be instructed to perform the same exercises before and after breakfast, lunch and dinner during the 4-week intervention period.

Placebo: abdominal and thoracic perimeter will be recorded but not shown to the patient and a pill of placebo containing 0.5 g glucose will be administered; patients will be instructed to take a pill of placebo before breakfast, lunch and dinner during the 4-week intervention period.

Primary Outcome Measure:

Number of rumination events measured by electromyography in response to the challenge meal before and after treatment.

Secondary Outcome Measures:

* Number of self perceived rumination events measured by questionnaires administered daily for 10 days will before and after treatment.
* Associated abdominal symptom measured by questionnaires administered daily for 10 days before and after treatment.
* Follow up: number of self perceived rumination events measured at 1, 3 and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Rumination syndrome

Exclusion Criteria:

* Relevant organic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Number of rumination events after a challenge meal measured by electromyography | 4 weeks
  Rumination events will be identified by recording the activity of the thoraco abdominal muscles (intercostals, external oblique, internal oblique, upper rectus, lower rectus) by electromyography after a challenge meal. The response to the meal will be measured before and after treatment.

SECONDARY OUTCOMES:
Number of self perceived rumination events. | 4 weeks
  Number of rumination events measured by questionnaires administered daily for 10 days before and after treatment.
Abdominal discomfort. | 4 weeks
  Abdominal discomfort will be measured by scales graded from 0 (no discomfort) to 10 (severe discomfort) administered daily for 10 days before and after treatment.
Number of self perceived rumination events up to 6 months. | up to 6 months
  Number of self perceived rumination events measured daily for 10 days using questionnaires at 1 month, 3 months and 6 months after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Vall d'Hebron Research Institute, Barcelona, Spain